CLINICAL TRIAL: NCT00733200
Title: Surgical Treatment of Hilar Cholangiocarcinoma: Minor or Major Liver Resection?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Ministry of Health, China (Other Government); Hepatic Surgery Clinical Research Centre of Hubei, China (Unknown)
Other Study IDs: chenxp002
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2008-08

CONDITIONS: Cholangiocarcinoma; Surgical Treatment; Hepatectomy
Keywords: Minor Liver Resection; Major Liver Resection; Hilar
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Nuclear Receptor Subfamily 4, Group A, Member 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Control group (No Intervention)
  Interventions: Procedure: Minor or Major Liver Resection

INTERVENTIONS:
Procedure: Minor or Major Liver Resection

SUMMARY:
The investigators conducted a prospective study to determine the safety and efficacy of minor and major hepatectomy selected by predetermined criteria in 138 patients with hilar cholangiocarcinoma. In selected patients, minor liver resection was a good treatment.

DETAILED DESCRIPTION:
Objective: To determine the safety and efficacy of minor and major hepatectomy selected by predetermined criteria in patients with hilar cholangiocarcinoma (HC).

Summary Background Data: For HC treated with hepatectomy, the extent of liver resection remains controversial despite extensive studies.

Methods: From January 2000 to December 2007, we prospectively studied patients who received surgical treatment for HC. Of the 187 patients who were surgically treated, 138 (73.8%) underwent resection with a curative intent. Minor hepatectomy was carried out in 93 patients who had Bismuth-Corlette types I, II and III HC without hepatic artery/portal vein invasion; and major hepatectomy in 45 patients who had type III HC with hepatic artery/portal vein invasion, or type IV HC.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for resectability were absence of peritoneal or liver metastases, tumor extension to beyond secondary biliary branches bilaterally, tumor extension to secondary portal venous branches bilaterally

Exclusion Criteria:

* not in accordance with the above criteria

Ages: 26 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
On multivariate analysis, prognostic factors significantly impacted on long-term survival were UICC tumor stage and histopathologic grade.